CLINICAL TRIAL: NCT05748483
Title: A Randomized, Double-Blind, Parallel-Group, Active Controlled Trial With Open-Label Safety Extension to Evaluate the Tolerability, Safety, and Efficacy of Atogepant Versus Topiramate in Subjects Requiring Preventive Treatment of Migraine (TEMPLE)
Brief Title: Comparative Study of Oral Atogepant Versus Oral Topiramate to Assess Adverse Events in Adult Participants With Migraine
Acronym: ATO-TOPIRAMATE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M22-061; 2022-501172-25-00 (Other: EU CT)
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Migraine
Keywords: Migraine; Episodic migraine; Chronic migraine; Atogepant; Topiramine; QULIPTA; Migraine prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atogepant (Experimental): Participants will receive atogepant in double-blind period. From Week 25, eligible participants will receive atogepant in open-label period.
  Interventions: Drug: Atogepant; Drug: Placebo for Topiramate
- Topiramate (Active Comparator): Participants will receive topiramate in double-blind period. From Week 25, eligible participants will receive atogepant in open-label period.
  Interventions: Drug: Atogepant; Drug: Placebo for Atogepant; Drug: Topiramate

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: QULIPTA
Drug: Placebo for Atogepant — Oral Tablet
  Arms: Topiramate
Drug: Topiramate — Oral Capsule
  Arms: Topiramate
Drug: Placebo for Topiramate — Oral Capsule
  Arms: Atogepant

SUMMARY:
A migraine is a moderate to severe headache on one side of the head that may be accompanied by throbbing, nausea, vomiting, sensitivity to light and sound, or other symptoms. The main goal of the study is to evaluate the tolerability (how patients handle the study treatment) and safety of atogepant compared to topiramate in participants with migraine.

Atogepant is a medicine currently approved for the preventive treatment of adult patients with episodic migraine (0 to 14 migraine days per month) and is being studied for the preventative treatment of migraine globally. Topiramate is an approved medication for migraine prevention. This study is conducted in 2 periods. In Period 1, participants will be randomly put into 1 of 2 groups at the start of the study to receive atogepant or topiramate. In Period 2, eligible participants will receive atogepant. Approximately 520 participants aged 18 and older will be enrolled in this study in approximately 85 sites across the world.

Participants will receive atogepant (and placebo for topiramate) or topiramate (and placebo for atogepant) for 24 weeks in Period 1. Both atogepant and placebo for atogepant are given as a tablet to take by mouth while topiramate and placebo for topiramate are given as a capsule to take by mouth. After 24 weeks, all eligible participants will receive atogepant for 52 weeks in Period 2. Participants are monitored for safety for 4 weeks after their last study treatment.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The safety and tolerability of the treatment will be checked by medical assessments, blood tests, checking for adverse events and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of migraine (with or without aura) for >= 12 months prior to screening (Visit 1).
* History of >= 4 migraine days per month who require preventive treatment of migraine and are eligible for conventional migraine prophylaxis.

Exclusion Criteria:

* Have used topiramate or atogepant in the past.
* Have clinically significant cardiovascular, cerebrovascular, hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Discontinued Treatment due to Adverse Events (AEs) | Up to Week 24 (Double-blind treatment period)
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Percentage of Participants Achieving >= 50% Improvement (Reduction) in Mean Monthly Migraine Days Based on mITT Population. | Month 4 to Month 6 (Double-blind treatment period)
  Improvement in mean monthly migraine days will be assessed.
Change From Baseline in Mean Monthly Migraine Days | Month 4 to Month 6 (Double-blind treatment period)
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.
Change from Baseline in HIT-6 (Headache Impact Test) Total Score | At Week 24
  The HIT-6 is a self-report questionnaire designed to evaluate the impact of headache on quality of life. Responses are based on frequency using a 5-point scale ranging from "never" to "always." The HIT-6 total score (which ranges from 36 to 78) is the sum of the responses, each of which is assigned a score ranging from 6 points (never) to 13 points (always).
Change From Baseline in Migraine Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) Role Function-Restrictive Domain Score | At Week 24
  MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality of life impairments attributed to migraine in the past 4 weeks. It is divided into three domains: Role Function Restrictive, Role Function Preventive, and Emotional Function domain. Participants respond to items using a 6-point scale ranging from "none of the time" to "all of the time." Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores indicate better quality of life.
Percentage of Participants Achieving a Rating of "Much Better" or "Very Much Better" Assessed by the Patient Global Impression of Change (PGIC) | At Week 24
  The PGIC is a single item used to measure the participants impression of overall change in migraine since the first dose of study medication. The measure uses a 7-point rating scale with responses ranging from "very much better" to "very much worse."
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function -Abilities Subset -Short Form 6a Version 2.0 score. | At Week 6
  The Patient Reported Outcomes Measurement Information System (PROMIS®) Cognitive Function and Cognitive Function Abilities Subset item banks assess participant perceived cognitive deficits. Facets include mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in these cognitive functions. The extent to which cognitive impairments interfere with daily functioning, whether other people observe cognitive impairments, and the impact of cognitive dysfunction on quality of life are also assessed. (Subset of participants when and where available)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (81):
- Austria (3):
  - Medizinische Universitaet Innsbruck /ID# 247213, Innsbruck, Tyrol
  - Konventhospital Barmherzige Brueder Linz /ID# 247217, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 247119, Vienna, Vienna
- Belgium (5):
  - Universitair Ziekenhuis Brussel /ID# 246959, Jette, Brussels Capital
  - Jessa Ziekenhuis /ID# 246954, Hasselt, Limburg
  - UZ Gent /ID# 246957, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan Brugge /ID# 246962, Bruges
  - CHR de la Citadelle /ID# 246964, Liège
- Canada (3):
  - Vancouver Island Health Authority /ID# 247733, Victoria, British Columbia
  - Maritime Neurology /ID# 247728, Halifax, Nova Scotia
  - Aggarwal and Associates Limited /ID# 247727, Brampton, Ontario
- Czechia (9):
  - CCR Ostrava, s.r.o. /ID# 245924, Ostrava, Ostrava-mesto
  - A-Shine s.r.o. /ID# 245923, Pilsen, Plzeň Region
  - Praglandia /ID# 247511, Prague, Praha 5
  - NeuroHK s.r.o. /ID# 247500, Hradec Králové
  - Pratia Pardubice a.s. /ID# 249017, Pardubice
  - Clintrial s.r.o. /ID# 245926, Prague
  - Pratia Prague s.r.o. /ID# 245925, Prague
  - Fakultni Thomayerova nemocnice /ID# 249016, Prague
  - INEP medical s.r.o. /ID# 245927, Prague
- France (3):
  - Hospices Civils de Lyon (HCL) - Hopital Louis Pradel /ID# 247562, Bron, Rhone
  - CHU Clermont Ferrand - Hopital Gabriel Montpied /ID# 247561, Clermont-Ferrand
  - AP-HP - Groupe Hospitalier 10e - Hopital Lariboisiere /ID# 249244, Paris
- Germany (25):
  - Studienzentrum fuer Neurologie und Psychiatrie /ID# 249236, Böblingen, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 246043, Tübingen, Baden-Wurttemberg
  - Neuropoint GmbH /ID# 246038, Ulm, Baden-Wurttemberg
  - Neuropraxis Muenchen Sued /ID# 246045, Unterhaching, Bavaria
  - Gesundheitszentrum Hoppegarten /ID# 249242, Hoppegarten, Brandenburg
  - Praxis fuer Neurologie, Psychiatrie und Psychotherapie /ID# 248427, Bad Homburg, Hesse
  - Kopfschmerzzentrum - Frankfurt /ID# 248686, Frankfurt am Main, Hesse
  - Klinische Forschung Hannover-Mitte GmbH /ID# 248565, Hanover, Lower Saxony
  - Studienzentrum Nord-West /ID# 246039, Westerstede, Lower Saxony
  - Klinische Forschung Schwerin GmbH /ID# 248074, Schwerin, Mecklenburg-Vorpommern
  - ZNS Siegen /ID# 251180, Siegen, North Rhine-Westphalia
  - Krankenhaus der Barmherzigen Brüder Trier /ID# 248564, Trier, Rhineland-Palatinate
  - Pharmakologisches Studienzentrum Chemnitz GmbH /ID# 246030, Chemnitz, Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 246040, Dresden, Saxony
  - Ambenet Hausarztpraxis /ID# 246028, Leipzig, Saxony
  - Schmerzklinik Kiel /ID# 246037, Kiel, Schleswig-Holstein
  - Neurologisches Facharztzentrum Berlin /ID# 248064, Berlin
  - Charite Universitaetsklinikum Berlin - Campus Virchow /ID# 246029, Berlin
  - NeuroZentrum Bielefeld /ID# 250758, Bielefeld
  - Neuro Centrum Odenwald /ID# 248067, Erbach im Odenwald
  - Universitaetsklinikum Essen /ID# 246033, Essen
  - Universitaetsmedizin Greifswald /ID# 248574, Greifswald
  - Klinische Forschung Hamburg GmbH /ID# 248620, Hamburg
  - Neurologische Gemeinschaftspraxis Kassel und Vellmar /ID# 248085, Kassel
  - Lewis Neurologie /ID# 250498, Stuttgart
- Hungary (5):
  - MIND Clinic /ID# 247867, Budapest
  - Clinexpert Kft /ID# 247868, Budapest
  - Semmelweis Egyetem /ID# 248428, Budapest
  - S-Medicon Kft /ID# 247682, Budapest
  - Debreceni Egeszsegugyi Kozpontja /ID# 247549, Debrecen
- Israel (4):
  - Meir Medical Center /ID# 247261, Kfar Saba, Central District
  - Hillel Yaffe Medical Center /ID# 247258, Hadera, H_efa
  - Shaare Zedek Medical Center /ID# 247259, Jerusalem, Jerusalem
  - Soroka University Medical Center /ID# 247260, Beersheba, Southern District
- Italy (6):
  - Azienda Ospedaliero Universitaria Careggi /ID# 247575, Florence, Firenze
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 247576, Naples, Napoli
  - IRCCS San Raffaele /ID# 247573, Rome, Roma
  - Azienda Ospedaliero-Universitaria di Modena /ID# 247578, Modena
  - Fondazione Mondino Istituto Neurologico Nazionale a Carattere Scientifico IRCCS /ID# 247579, Pavia
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 247580, Roma
- Poland (9):
  - Solumed Centrum Medyczne /ID# 247317, Poznan, Greater Poland Voivodeship
  - Clinical Research Center Sp. z.o.o. Medic-R sp. k /ID# 247323, Poznan, Greater Poland Voivodeship
  - Vitamed Galaj i Cichomski Sp.j. /ID# 247314, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Athleticomed Sp. z o.o /ID# 250790, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Instytut Zdrowia Dr Boczarska Jedynak /ID# 247315, Oświęcim, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 247298, Lublin, Lublin Voivodeship
  - RCMed Oddzial Sochaczew /ID# 247378, Sochaczew, Masovian Voivodeship
  - ETG Neuroscience Sp. z o.o. /ID# 247331, Warsaw, Masovian Voivodeship
  - Silmedic Sp. z o.o. /ID# 247376, Katowice, Silesian Voivodeship
- Portugal (6):
  - Hospital Garcia de Orta /ID# 247163, Almada, Setúbal District
  - 2CA-Braga, Hospital de Braga /ID# 247165, Braga
  - Hospital da Luz Lisboa /ID# 247168, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 247167, Lisbon
  - Hospital Prof. Doutor Fernando Fonseca, EPE /ID# 247172, Lisbon
  - Unidade Local de Saúde de Matosinhos, EPE /ID# 247169, Matosinhos Municipality
- United Kingdom (3):
  - The Adam Practice /ID# 248880, Poole, Dorset
  - Duplicate_NHS Greater Glasgow and Clyde /ID# 247979, Glasgow, Scotland
  - West Walk Surgery /ID# 252855, Bristol

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-061